CLINICAL TRIAL: NCT04268901
Title: Effectiveness of Virtual Reality to Reduce Pain/Anxiety During Routine Painful Procedures
Brief Title: VR to Reduce Pain/Anxiety During Painful Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: AppliedVR Inc. (Industry)
Responsible Party: Principal Investigator, Jeffrey I Gold, PhD, Professor of Anesthesiology, Pediatrics, and Psychiatry & Behavioral Sciences, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHLA-15-00549
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Phlebotomy; Orthopedics; Radiology; Pain; Anxiety; Virtual Reality; Allergy; Gastroenterology
Keywords: phlebotomy; radiology; orthopedics; infusion; IV stick; cast removal; pain; anxiety; virtual reality; allergy; gastroenterology; anorectal manometry
MeSH Terms: conditions — Pain; Anxiety Disorders; Hypersensitivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard of Care (No VR) Randomization (No Intervention): In the standard of care treatment condition, participants will receive the standard CHLA treatment protocol for the medical procedure.
- VR Randomization (Experimental): Children in the VR condition will undergo the invasive procedure while distracted by interaction with an immersive virtual environment (VE) presented via a head mounted display (HMD). The intervention group will receive standard CHLA treatment with VR distraction.
  Interventions: Device: Samsung Gear VR; Device: Merge VR; Device: Oculus Go

INTERVENTIONS:
Device: Samsung Gear VR — Participants 13 -21 years old can use the Samsung Gear VR. The VE to be used in this study is mobile based (Samsung with the Gear VR) and has active matrix LCDs with high pixel resolution, creating a bright, vibrant color and a quality image. The VR game is equipped with a head-tracking system, enabling the player to look around the virtual environment. In addition, there is the option to interact with the VR environment using a tap pad located on the side of the helmet. Therefore, the child will be receiving distraction via 3-D visual and auditory sensory, and tactile feedback, thus supplying a multi-sensory immersive experience. While wearing these glasses, the children only can see the HMD screen so that the immersion and presence will be increased. The VR glasses will be sanitized before every use so that the chance of infection will be minimized.
  Arms: VR Randomization
Device: Merge VR — Participants 10-21 years can use the Merge. The VE to be used in this study is mobile based (Pixel with the Merge) and has active matrix LCDs with high pixel resolution, creating a bright, vibrant color and a quality image. The VR game is equipped with a head-tracking system, enabling the player to look around the virtual environment. In addition, there is the option to interact with the VR environment using a tap pad located on the side of the helmet. Therefore, the child will be receiving distraction via 3-D visual and auditory sensory, and tactile feedback, thus supplying a multi-sensory immersive experience. While wearing these glasses, the children only can see the HMD screen so that the immersion and presence will be increased. The VR glasses will be sanitized before every use so that the chance of infection will be minimized.
  Arms: VR Randomization
Device: Oculus Go — Participants 7-21 years can use the Oculus Go. The visual a bright, vibrant color and a quality image. The VR game is equipped with a head-tracking system, enabling the player to look around the virtual environment. In addition, there is the option to interact with the VR environment using a handheld remote. Therefore, the child will be receiving distraction via 3-D visual and auditory sensory, and tactile feedback, thus supplying a multi-sensory immersive experience. While wearing these glasses, the children only can see the HMD screen so that the immersion and presence will be increased. The VR glasses will be sanitized before every use so that the chance of infection will be minimized.
  Arms: VR Randomization

SUMMARY:
This study aims to test the effectiveness of virtual reality (VR) as a non-pharmaceutical intervention to reduce pain and anxiety in children undergoing painful procedures in Phlebotomy, Radiology, Infusion, Orthopedics, Gastroenterology, and Immunology, amongst others, at CHLA, as measured by self- and proxy-report. Examples of the painful procedures include IV sticks, cast removals, allergy testing, and anorectal manometries.

DETAILED DESCRIPTION:
Distraction is a form of non pharmacological intervention for reducing pain and anxiety in children during painful medical procedures (e.g., venipuncture, IV placement). Recent technological developments in the area of virtual reality (VR) provide new and potentially more effective ways of distracting children from the pain and anxiety associated with medical procedures. While initial studies of VR pain distraction are promising, few have studied the effectiveness of the technology in children, using a multi-method approach. The current study aims to recruit 240 children ages 7-21 and their caregivers who arrive at the hospital for an outpatient painful medical procedure. Children and their parents will be randomly assigned to one of two treatment conditions: 1) existing hospital standard of care or 2) standard of care plus distraction via VR. Children and caregivers will be asked to complete measures assessing pain and anxiety both before and after the procedure. In addition, objective measures of child pain and distress during the medical procedure will be taken using coding of behavioral/verbal expressions. Univariate Analysis of Variance (ANOVA) will be used to compare differences in primary and secondary outcome variables in VR + standard of care to standard of care only conditions when pre and post-operative measures are available. Univariate ANOVA will be used to compare conditions on post-operative variables.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Children:

1. Children who are 7-21 years old
2. Children who are English speaking (caregivers may be Spanish English speaking or Spanish speaking)
3. Children who are undergoing a painful medical procedure (e.g., venipuncture, IV placement, PICC lines, wound care, cast removal, botox injections) are eligible to participate in this project.
4. Only children who are in the normal range of development will be recruited for this study. This will be assessed by report from the parents. The rationale for excluding patients with developmental delay is that due to their cognitive impairments, such children react to the stressors of surgery differently than do children without such developmental delay. It is unclear how such children would use the interventions included in this study, and it is likely that their responses on baseline and outcome measures will differ from children of normal developmental parameters.

Inclusion criteria for healthcare providers:

1. Healthcare providers must be 18 years old or older
2. Healthcare providers must be Children's Hospital Los Angeles staff
3. Healthcare providers may participate if they have witnessed and/or administered the medical procedure

Exclusion Criteria:

1. Children who are currently taking pain medication or anxiolytic medication will be excluded from this study.
2. Children with a psychiatric disorder, organic brain syndrome, mental retardation, or other known cognitive/neurological disorders
3. Children with visual, auditory, or tactile deficits that would interfere with the ability to complete the experimental tasks
4. Children with a history of seizure disorder.
5. Children currently sick with flu-like symptoms or experiencing a headache or earache.
6. Children with known or suspected motion sickness

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 700 (Estimated)
Dates: Start 2016-02-19 (Actual); Primary Completion 2025-12-06 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
VAS | Approximately 5 minutes to one hour before procedure
  VAS anticipatory anxiety measure: The VAS anticipatory anxiety measure is a vertical VAS, anchored with 0 at the bottom indicating the least amount and 10 at the top indicating the greatest amount, in response to the instruction to rate "how nervous, afraid, or worried" they were about the upcoming task. The scale also has color cues, graded from yellow at the bottom to dark red at the top, as well as a neutral face at the bottom and a face showing a negative expression at the top. Prior research used the VAS to rate anticipatory anxiety and pain in children.
Faces Pain Scale (FPS-R) | Approximately 5 minutes to one hour before procedure
  Revised is an updated version of the Wong-Baker Faces Pain Rating Scale depicting no pain as a neutral expression as compared with the smiling face of the original measure. The child is asked to point to the face cartoon that depicts how they are currently feeling because of their pain. Face measures are thought to measure pain intensity, and the Wong-Baker Faces measure has demonstrated good reliability and validity.
Facial Affective Scale | Approximately 5 minutes to one hour before procedure
  A faces scale to predict pediatric pain unpleasantness.
Child State Anxiety Index (CASI) or Anxiety Sensitivity Index (ASI) if 18 and older | Approximately 5 minutes to one hour before procedure
  CASI is an 18-item scale that measures the tendency to view anxiety-related bodily sensations as dangerous (e.g., ''It scares me when my heart beats fast''). Items are scored on a 3-point scale (none, some, a lot), and total scores are calculated by summing all items. The CASI has demonstrated high internal consistency and adequate test-retest reliability. The CASI correlates well with measures of trait anxiety but also accounts for variance in fear not attributable to trait anxiety measures
Malaise Scale | Approximately 5 minutes to one hour before procedure
  The MS is a six-point scale indicating level of nausea from (1) no symptoms to (6) being sick The MS is completed before and after administration of the VR game to monitor for any signs of nausea. Instructions to the child are as follows: "This is a scale from one to six. One means that you feel fine and no different to how you normally feel. Two means that you feel a little bit different or funny but not sick in the tummy. Three means that you feel a little bit sick and four means that you feel more than a little bit sick but not really sick. Five means that you feel really sick, like you are going to throw up or vomit and six means that you are being sick or vomiting. I'm going to ask you every few minutes how you feel. I want you to tell me which number from one to six best describes how you feel at that time."
Child Presence Questionnaire | Approximately 5-15 minutes after procedure
  The Child Presence Questionnaire was developed out of a content analysis of the entire domain of adult presence items and selection and adaptation of appropriate items for assessing the child's sense of believability of their experience. This 16-item measure is verbally administered to children and asks them to respond according to a 3-point Likert-like format. Items assess the child's sense of involvement, realism, and transportation into the experience. Patients in the VR condition will complete the Child Presence Questionnaire post-procedure to assess level of VR immersion.
Child Satisfaction Survey | Approximately 5-15 minutes after procedure
  The child survey is 13-item, Likert-like survey to assess child estimates of pain reduction, fear reduction, decreased behavioral distress, and overall satisfaction; it mirrors the parent survey. There are two versions, one for each treatment condition. Two versions of the survey exist, to account for condition (VR vs. standard of care).
Parent Satisfaction Survey | Approximately 5-15 minutes after procedure
  The parent survey is 16-item, Likert-like survey to assess parent estimates of pain reduction, fear reduction, decreased behavioral distress, and overall satisfaction. Two versions of the survey exist, to account for condition (VR vs. standard of care).
Healthcare Provider Survey | Approximately 5-15 minutes after procedure
  The healthcare provider survey is a 7-item Likert-like investigator-developed survey to assess their estimates of pain and anxiety management, cooperation, and satisfaction with the procedure. Healthcare providers are also invited to write comments about the use of VR (if applicable) during the IV placement procedure.
VAS | Approximately 5-15 minutes after procedure
  VAS anticipatory anxiety measure: The VAS anticipatory anxiety measure is a vertical VAS, anchored with 0 at the bottom indicating the least amount and 10 at the top indicating the greatest amount, in response to the instruction to rate "how nervous, afraid, or worried" they were about the upcoming task. The scale also has color cues, graded from yellow at the bottom to dark red at the top, as well as a neutral face at the bottom and a face showing a negative expression at the top. Prior research used the VAS to rate anticipatory anxiety and pain in children.
Faces Pain Scale (FPS-R) | Approximately 5-15 minutes after procedure
  Revised is an updated version of the Wong-Baker Faces Pain Rating Scale depicting no pain as a neutral expression as compared with the smiling face of the original measure. The child is asked to point to the face cartoon that depicts how they are currently feeling because of their pain. Face measures are thought to measure pain intensity, and the Wong-Baker Faces measure has demonstrated good reliability and validity.
Facial Affective Scale | Approximately 5-15 minutes after procedure
  A faces scale to predict pediatric pain unpleasantness.
Malaise Scale | Approximately 5-15 minutes after procedure
  The MS is a six-point scale indicating level of nausea from (1) no symptoms to (6) being sick The MS is completed before and after administration of the VR game to monitor for any signs of nausea. Instructions to the child are as follows: "This is a scale from one to six. One means that you feel fine and no different to how you normally feel. Two means that you feel a little bit different or funny but not sick in the tummy. Three means that you feel a little bit sick and four means that you feel more than a little bit sick but not really sick. Five means that you feel really sick, like you are going to throw up or vomit and six means that you are being sick or vomiting. I'm going to ask you every few minutes how you feel. I want you to tell me which number from one to six best describes how you feel at that time."

SECONDARY OUTCOMES:
CAMPIS-R | Peri-procedure
  The CAMPIS-R is a standardized rating scale that codes videotaped verbal interactions in the pediatric treatment room. The CAMPIS-R codes the subject, speaker, phase of medical procedure, verbal content, affective tone, and to whom vocalizations are directed. Adult vocalizations are coded as coping-promoting (nonprocedural talk or humor directed to the child, commands to engage in coping strategies), distress-promoting (reassuring comments, apologies, giving control to the child, criticism, and empathetic statements), or neutral (humor to adults, nonprocedural talk to adults, child's condition talk, commands for procedural activity, praise, notification of procedure to come, behavioral commands to child, checking child's status). Two independent study team coders will complete the CAMPIS-R while reviewing the videotape from each of the I&D of abscess procedures.

OTHER OUTCOMES:
Demographic Survey | Approximately 5 minutes to one hour before procedure
  A brief demographic survey will be administered to parent regarding their child's age, ethnicity, grade in school, and any medical conditions or learning problems they may have.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey I Gold, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rothbaum BO, Hodges L, Kooper R. Virtual reality exposure therapy. J Psychother Pract Res. 1997 Summer;6(3):219-26. PMID 9185067
- [Background] Schneider SM, Workman ML. Effects of virtual reality on symptom distress in children receiving chemotherapy. Cyberpsychol Behav. 1999;2(2):125-34. doi: 10.1089/cpb.1999.2.125. PMID 19178248
- [Background] Riva G, Bacchetta M, Baruffi M, Rinaldi S, Molinari E. Experiential cognitive therapy: a VR based approach for the assessment and treatment of eating disorders. Stud Health Technol Inform. 1998;58:120-35. PMID 10350912
- [Background] Stanton, D., Foreman, N., Wilson, P., & Duffy, H. (2002). Use of virtual environments to acquire spatial understanding of real world multi-level environments. 13-19. Paper presented at Fourth International Conference on Disability, Virtual Reality and Associated Technologies (ICDVRAT), Vesprem, Hungary.
- [Background] Parsons TD, Bowerly T, Buckwalter JG, Rizzo AA. A controlled clinical comparison of attention performance in children with ADHD in a virtual reality classroom compared to standard neuropsychological methods. Child Neuropsychol. 2007 Jul;13(4):363-81. doi: 10.1080/13825580600943473. PMID 17564852
- [Background] McComas, J., Pivik, J., & Laflamme, M. (1998). Children's transfer of spatial learning from virtual reality to real environments. CyberPsychology & Behavior, 1(2), 121-128. https://doi.org/10.1089/cpb.1998.1.121
- [Background] Pugnetti L, Mendozzi L, Barbieri E, Motta A. VR experience with neurological patients: basic cost/benefit issues. Stud Health Technol Inform. 1998;58:243-8. PMID 10350925
- [Background] Hoffman HG, Patterson DR, Carrougher GJ, Sharar SR. Effectiveness of virtual reality-based pain control with multiple treatments. Clin J Pain. 2001 Sep;17(3):229-35. doi: 10.1097/00002508-200109000-00007. PMID 11587113
- [Background] Mahrer NE, Gold JI. The use of virtual reality for pain control: a review. Curr Pain Headache Rep. 2009 Apr;13(2):100-9. doi: 10.1007/s11916-009-0019-8. PMID 19272275
- [Background] Malloy KM, Milling LS. The effectiveness of virtual reality distraction for pain reduction: a systematic review. Clin Psychol Rev. 2010 Dec;30(8):1011-8. doi: 10.1016/j.cpr.2010.07.001. Epub 2010 Jul 13. PMID 20691523
- [Background] Birnie KA, Noel M, Parker JA, Chambers CT, Uman LS, Kisely SR, McGrath PJ. Systematic review and meta-analysis of distraction and hypnosis for needle-related pain and distress in children and adolescents. J Pediatr Psychol. 2014 Sep;39(8):783-808. doi: 10.1093/jpepsy/jsu029. Epub 2014 Jun 2. PMID 24891439
- [Background] Cohen LL, Rodrigues NP, Lim CS, Bearden DJ, Welkom JS, Joffe NE, McGrath PJ, Cousins LA. Automated parent-training for preschooler immunization pain relief: a randomized controlled trial. J Pediatr Psychol. 2015 Jun;40(5):526-34. doi: 10.1093/jpepsy/jsu162. Epub 2015 Jan 30. PMID 25638483
- [Background] MacLaren JE, Cohen LL. A comparison of distraction strategies for venipuncture distress in children. J Pediatr Psychol. 2005 Jul-Aug;30(5):387-96. doi: 10.1093/jpepsy/jsi062. Epub 2005 Feb 23. PMID 15944166
- [Background] Taddio A, Goldbach M, Ipp M, Stevens B, Koren G. Effect of neonatal circumcision on pain responses during vaccination in boys. Lancet. 1995 Feb 4;345(8945):291-2. doi: 10.1016/s0140-6736(95)90278-3. PMID 7837863
- [Background] Fradet C, McGrath PJ, Kay J, Adams S, Luke B. A prospective survey of reactions to blood tests by children and adolescents. Pain. 1990 Jan;40(1):53-60. doi: 10.1016/0304-3959(90)91050-S. PMID 2339016
- [Background] Van Cleve L, Johnson L, Pothier P. Pain responses of hospitalized infants and children to venipuncture and intravenous cannulation. J Pediatr Nurs. 1996 Jun;11(3):161-8. doi: 10.1016/S0882-5963(96)80049-2. PMID 8667153
- [Background] Hoffman HG, Garcia-Palacios A, Patterson DR, Jensen M, Furness T 3rd, Ammons WF Jr. The effectiveness of virtual reality for dental pain control: a case study. Cyberpsychol Behav. 2001 Aug;4(4):527-35. doi: 10.1089/109493101750527088. PMID 11708732
- [Background] Hoffman, H. G., Patterson, D. R., Carrougher, G. J., Nakamura, D., Moore, M., Garcia-Palacios, A., & Furness, T. A. III. (2001). The effectiveness of virtual reality pain control with multiple treatments of longer durations: A case study. International Journal of Human-Computer Interaction, 13(1), 1-12. https://doi.org/10.1207/S15327590IJHC1301_1
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Gershon J, Zimand E, Pickering M, Rothbaum BO, Hodges L. A pilot and feasibility study of virtual reality as a distraction for children with cancer. J Am Acad Child Adolesc Psychiatry. 2004 Oct;43(10):1243-9. doi: 10.1097/01.chi.0000135621.23145.05. PMID 15381891
- [Background] Windich-Biermeier A, Sjoberg I, Dale JC, Eshelman D, Guzzetta CE. Effects of distraction on pain, fear, and distress during venous port access and venipuncture in children and adolescents with cancer. J Pediatr Oncol Nurs. 2007 Jan-Feb;24(1):8-19. doi: 10.1177/1043454206296018. PMID 17185397
- [Derived] Gold JI, Akbar KM, Avila S, Ngo NH, Klein MJ. Exploring Relations Between Unique Patient Characteristics and Virtual Reality Immersion Level on Anxiety and Pain in Patients Undergoing Venipuncture: Secondary Analysis of a Randomized Control Trial. J Med Internet Res. 2024 Jul 1;26:e53196. doi: 10.2196/53196. PMID 38949862